CLINICAL TRIAL: NCT00257478
Title: A Study for the Treatment of Hormone Refractory Prostate Cancer (HRPC) in Patients Previously Treated With Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 155-CL-007
Record Dates: First submitted 2005-11-22; First posted 2005-11-23 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Prostate Cancer; Cancer of Prostate; Prostatic Cancer; Cancer of the Prostate
Keywords: Treatment Efficacy; Treatment Effectiveness; Disease Management; Treatment; Safety
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sepantronium

INTERVENTIONS:
Drug: YM155

SUMMARY:
A study for the treatment of hormone refractory prostate cancer (HRPC) in patients previously treated with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed prostate cancer.
* Prior chemotherapy regimen for prostate cancer

Exclusion Criteria:

* History of other malignancy in the last 5 years
* Major surgery within the past 21 days

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: D. Buell, MD, Study Director — Astellas Pharma US, Inc.
Locations (9):
- United States (7):
  - Tuscon, Arizona
  - Los Angeles, California
  - Coeur d'Alene, Idaho
  - New York, New York
  - The Bronx, New York
  - Philadelphia, Pennsylvania
  - San Antonio, Texas
- Amsterdam, Netherlands
- Sutton, Surry, United Kingdom